CLINICAL TRIAL: NCT03579914
Title: Combined Metoprolol and Remote Ischemic Conditioning in Cardioprotection of Anterior ST-segment Elevation Myocardial Infarction (METRICATION)
Brief Title: Effect of Intravenous Metoprolol Combining RIC on Myocardial Protection in STEMI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Yu Bo, director, Harbin Medical University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1301102
Record Dates: First submitted 2018-05-17; First posted 2018-07-09 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Anterior Myocardial Infarction; Heart Failure
Keywords: Anterior Myocardial Infarction; Intravenous Metoprolol; RIC; Myocardial Protection
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; Heart Failure | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo group (Placebo Comparator): Patients receive intravenous placebo injection.
  Interventions: Drug: intravenous Placebo
- Intravenous metoprolol group (Experimental): Patients receive intravenous metoprolol injection.
  Interventions: Drug: Metoprolol Injectable Product
- RIC group (Experimental): Patients receive RIC treatment.
  Interventions: Device: Romote Ischemic Conditioning (RIC)
- Intravenous metoprolol and RIC group (Experimental): Patients receive intravenous metoprolol injection and RIC treatment.
  Interventions: Combination Product: Metoprolol & RIC

INTERVENTIONS:
Drug: intravenous Placebo — Patients receive intravenous Placebo (saline) injection
  Arms: Placebo group
Drug: Metoprolol Injectable Product — Patients receive intravenous Metoprolol injection
  Arms: Intravenous metoprolol group
Device: Romote Ischemic Conditioning (RIC) — Patients receive RIC treatment
  Arms: RIC group
Combination Product: Metoprolol & RIC — Patients receive Metoprolol & RIC treatment
  Arms: Intravenous metoprolol and RIC group

SUMMARY:
The main purpose of this study is to compare the myocardial protection effect of intravenous metoprolol combined with remote ischemic conditioning (RIC) and single treatment before reperfusion in Chinese patients with anterior STEMI. This study sought to find possible strategies to further improve myocardial protection in Chinese patients with anterior STEMI.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized controlled study. It is planned to enroll 1200 patients with anterior STEMI. Immediately after the first medical contact, the patients who were determined by the investigator to meet the inclusion/exclusion criteria were randomized through the interactive web response system (IWRS) and received different pre-reperfusion treatments. The four groups were placebo group, metoprolol group, remote ischemic conditioning (RIC) group and metoprolol & RIC group. Subsequently, the investigator conduct diagnosis and treatment according to the patient's specific conditions and check the serum level of myocardial damage markers (i.e. CK and CK-MB) at the time of admission, 12, 24, 36, 48, 60 hours, respectively. If the patient undergoes PCI treatment, additional detection of myocardial damage markers immediately after PCI is also required. All patients were followed for 1 year with an office visit or a telephone call at 1, 3, 6, 9 and 12 months to evaluate the health status and adverse clinical events of patients.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18 to 80 years;
2. presenting within 12 h of symptoms onset, with anterior STEMI and planned for pPCI; anterior STEMI was defined as the occurrence of >20 min of chest pain and ST-segment elevation (>2 mm) in at least 2 contiguous precordial leads;
3. sign informed consent;

Exclusion Criteria:

1. systolic blood pressure < 110mmHg;
2. cardiogenic shock or with heart failure symptoms, Killip III~IV;
3. allergic history of metoprolol;
4. history of asthma or the need for bronchodilators;
5. PR interval > 240ms, II~III atrioventricular block；
6. heart rate < 60 beats/min;
7. unable to consent;
8. pregnancy and lactation women;
9. life expectancy for diseases (i.e. cancer) < 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1206 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct size | 60 hours
  Estimating myocardial infarct size by area under CK, CK-MB curve

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 1 year
  Composition of death, heart failure, reinfarction, revascularization, malignant ventricular arrhythmias, stroke)
Incidence of heart failure | 1 year
  Incidence of heart failure
myocardial infarct size measured by MRI (optional) | 7 days after AMI
  myocardial infarct size measured by MRI (optional)
Safety endpoint: incidence of severe bradycardia or hypotension | 24 hours
  Severe bradycardia (heart rate <40bpm) or hypotension (systolic blood pressure <80mmHg)

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Peking Univerisity People'Hospital, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Guangdong general hospital, Guangzhou, Guangdong
  - Second hospital of hebei medical university, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The first affiliated hospital of Zhengzhou medical university, Zhengzhou, Henan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - the second affiliated hospital of Dalian medical university, Dalian, Liaoning
  - Shenyang military district general hospital of the people's liberation army, Shenyang, Liaoning
  - The first affiliated hospital of military medical university, Xi’an, Shanxi
  - Third Military Medical University, Chongqing, Sichuan
  - The General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang